CLINICAL TRIAL: NCT01769794
Title: Chinese Medicinal Treatment on Mild Hand, Foot, and Mouth Disease: Multicenter, Prospective, Randomized Double-blind, Placebo-controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Chengdu University of Traditional Chinese Medicine (Other); Beijing Children's Hospital (Other); Tianjin infectious disease hospital (Unknown); Tangshan infectious disease hospital (Unknown); The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other); Tianjin Zhongshenghaitian Pharmaceutical Co. Ltd. (Unknown)
Responsible Party: Principal Investigator, Liyun He, chief, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ChinaACMS-HFMD
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: Hand, Foot and Mouth Disease; Medicine, Chinese Traditional; Enterovirus; Fever
MeSH Terms: conditions — Hand, Foot and Mouth Disease; Enterovirus Infections; Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Western therapy & Placebo (Active Comparator): Western therapy(oral care, skin care and reducing temperature) Placebo for JET(Jinlianqingre Effervescent Tablets )
  Interventions: Drug: Western therapy; Drug: Placebo(for JET)
- Western therapy & JET (Experimental): Jinlianqingre Effervescent Tablets plus western therapy
  Interventions: Drug: Western therapy; Drug: JET

INTERVENTIONS:
Drug: Western therapy — Physical cooling paste or warm bathing, vitamin B, vitamin C. On the basis of the attending physician's judgment, participants were allowed to use Ibuprofen suspension if their body temperature was greater than 38.5℃. Likewise, the need for antibiotics was determined by the attending physicians. The use of acetaminophen or antibiotics was recorded on the case record form
Drug: JET — 4g/tablet, One tablet each time (Taken after dissolved in 50ml boiled water, 3 times daily if body temperature≥38.5℃)
  Other Names: Jinlianqingre Effervescent Tablets
  Arms: Western therapy & JET
Drug: Placebo(for JET) — placebos prepared identical in color, taste and consistency to the JET (supplied by Zhongshenghaitian Pharmaceutical, Tianjin, China)
  Arms: Western therapy & Placebo

SUMMARY:
The study is aimed to evaluate the effectiveness and safety of Jinlianqingre Effervescent Tablets, a traditional Chinese medicine (TCM), in the treatment of Uncomplicated hand, foot, and mouth disease (HFMD).

DETAILED DESCRIPTION:
By adopting a multicenter, prospective, randomized double-blind, placebo-controlled, this study is aimed to evaluate the effectiveness, safety of a traditional Chinese medicine, Jinlianqingre Effervescent Tablets, for treatment Uncomplicated HFMD, and to provide scientific evidence for the construction of TCM methods in treating HFMD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild hand-foot-mouth disease patients according to Hand-Foot-Mouth Disease Treatment Guidelines 2010 issued by China's Ministry of Health;
* Within 48 hours of onset of fever and rash symptom.
* Age of 1-13 years.
* Documented body temperature 37.4 °C-39.0°C
* Patients or their guardians agree to participate in this study and signed the informed consent form.

Exclusion Criteria:

* Complicated with other serious diseases such as chronic hepatitis,chronic diarrhea disease,chronic diarrhea, congenital heart disease, acute or chronic nephritis and blood diseases.
* With history of allergies on traditional Chinese medicine.
* Attending other clinical studies on HFMD after diagnosed.

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 288 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The time of body temperature going back to normal | 10 days
  Referring to the time of the armpit temperature of lower than 37.0 degrees Celsius, lasting for at least 24 hours, after the medicine is taken.

SECONDARY OUTCOMES:
Healing time of skin or oral mucosa lesions symptom | 10 days
  Referring to the number of days in the total-contact cast until the skin completely closed after the medicine is used.
Score of skin or oral mucosa lesions symptom during the study period time | 10 days
  Referring to Symptoms were hands, feet, oral mucosa lesions, buttock, crissum, back and four limbs. Each symptom was scored as 0 (none), 1 (mild), 2 (modest), or 3 (severe).
the length of hospital stay | 10 days
major complications rate | 10 days
  Referring to pulmonary edema, cardiac damage, pneumonia, secondary infection, meningitis, encephalomyelitis et al.

CONTACTS AND LOCATIONS:
Overall Officials: Boyan Liu, chief physician, Study Chair — China Academy of Chinese Medical Sciences; Guoliang Zhang, chief, Study Chair — The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine
Locations (4):
- China (4):
  - Tangshan infectious disease hospital, Tangshan, Hebei
  - Affiliated Hospital of Chengdu university of Traditional Chinese Medicine, Chengdu, Sichuan
  - Beijing children's hospital, Beijing
  - Tianjin infectious disease hospital, Tianjin